CLINICAL TRIAL: NCT02361450
Title: Retrograde Colonic Irrigation to Manage Spina Bifida Functional Digestive Sequelae: a Multicenter, Prospective, Randomized Controlled Trial
Acronym: IRRICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-A01520-45
Record Dates: First submitted 2015-02-02; First posted 2015-02-11 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Spina Bifida
Keywords: Faecal incontinence; Spina Bifida; Enema; Constipation; Myelomeningocele; Human
MeSH Terms: conditions — Spinal Dysraphism; Encopresis; Constipation; Meningomyelocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Retrograde Colonic Irrigation with usual care (Experimental): In the experimental group, retrograde colonic irrigation sessions will be scheduled in addition to conventional treatment according to a progressive volume program.
  Interventions: Device: Retrograde Colonic Irrigation; Other: Usual Care
- Usual Care (Active Comparator): In the comparator group, patients will receive conventional care, according to each clinical center habits.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Retrograde Colonic Irrigation
  Arms: Retrograde Colonic Irrigation with usual care
Other: Usual Care

SUMMARY:
Spina Bifida is a developmental congenital disorder caused by the incomplete closing of the embryonic neural tube, leading to serious malformations of the nervous system. Caudal neuropore malformations almost always lead to sensory-motor deficits (including complete paraplegia) with orthopedic deformations, pressure sores, and pelvic/perineal neurological dysfunctions (affecting the bladder-sphincter, anorectal, and genital sphere).

The purpose of the study is to assess the efficacy of retrograde colonic irrigation associated with usual care (medical treatments, patient education) on anorectal dysfunction (incontinence and/or constipation), compared to usual care only.

DETAILED DESCRIPTION:
Sphincter dysfunctions impair the quality of life and patients' self-esteem. However, defecation disorders are important issues the Spina Bifida National Reference Center has to deal with. Indeed, more than half of patients are concerned. These disorders are mainly due to fecal stasis. Treatments include laxatives and hygiene recommendations. Colonic irrigation can also be useful, especially to achieve colonic vacuity and improve continence. The use of intra-rectal balloon inflation probes and the control of instillation flow improved retrograde colonic irrigation efficacy. Nevertheless, this technique is currently not evaluated in young adults suffering from Spina Bifida functional digestive sequelae, who are mainly concerned by Malone enema.

The purpose of the study is to assess the efficacy of retrograde colonic irrigation associated with usual care (medical treatments, patient education) on anorectal dysfunction (incontinence and/or constipation), compared to usual care only.

ELIGIBILITY:
Inclusion Criteria:

* Patients aging at least 15 years old with Spina Bifida neurological pelvi-perineal sequelae, objected by neurologic exam , functional urinary and/or anorectal and/or neurophysiological data,
* Patients with NBD score above 9,
* Written and informed consent (Minor children may be included with the consent of the two parents).

Exclusion Criteria:

* Patients with psychiatric disorders, cognitive or intellectual disabilities compromising the assessment of primary outcome measure,
* Patients using currently irrigation colonic technique,
* Patients with functional colostomy, known anal or colorectal stenosis, colorectal cancer, acute or chronic inflammatory disease, recent anal or colorectal surgery for less than 3 months, polyp removal for less than 4 weeks, ischemic colitis.
* Patients with urinary trophic or orthopedic disease with planned surgery during inclusion or follow-up periods,
* Patients with progressive anal disease (suppuration, hemorrhoid or rectal prolapse)
* Patient with a hard follow-up ( judged by the investigator)
* Person involved in another clinical trial
* Pregnant women
* Person with a measure of legal protection (guardianship)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Neurogenic Bowel Dysfunction (NBD) score | Ten weeks after inclusion

SECONDARY OUTCOMES:
Questionnaire data of incontinence and constipation (Cleveland scores) | Ten weeks after inclusion
Questionnaire data of incontinence and constipation (Cleveland scores) | Twenty-four weeks after inclusion
Quality of life | Ten weeks after inclusion
  Quality of life will be assess by semi-quantified scales
Quality of life | Twenty-four weeks after inclusion
  Quality of life will be assess by semi-quantified scales
Self esteem (Rosenberg scale) | Ten weeks after inclusion
Functional digestive score (NBD) | Twenty-four weeks after inclusion
Cumulative time spent using restrooms | Ten weeks after inclusion
  Cumulative time spent using restrooms will be collected with a patient reported outcome questionnaire
Cumulative time spent using restrooms | Twenty-four weeks after inclusion
  Cumulative time spent using restrooms will be collected with a patient reported outcome questionnaire
Number of accidents of incontinence | Ten weeks after inclusion
  Number of accidents of incontinence will be collected with a patient reported outcome questionnaire
Number of accidents of incontinence | Twenty-four weeks after inclusion
  Number of accidents of incontinence will be collected with a patient reported outcome questionnaire
Number of incontinence guards used | Ten weeks after inclusion
  Number of incontinence guards used will be collected with a patient reported outcome questionnaire
Number of incontinence guards used | Twenty-four weeks after inclusion
  Number of incontinence guards used will be collected with a patient reported outcome questionnaire
Type of incontinence guards used | Ten weeks after inclusion
  Type of incontinence guards (panty liner, pad, nappy) used will be collected with a patient reported outcome questionnaire
Type of incontinence guards used | Twenty-four weeks after inclusion
  Type of incontinence guards (panty liner, pad, nappy) used will be collected with a patient reported outcome questionnaire
Number of stools | Ten weeks after inclusion
  Number of stools will be collected with a patient reported outcome questionnaire
Number of stools | Twenty-four weeks after inclusion
  Number of stools will be collected with a patient reported outcome questionnaire
Stools consistency | Ten weeks after inclusion
  Stools consistency will be collected with a patient reported outcome questionnaire
Stools consistency | Twenty-four weeks after inclusion
  Stools consistency will be collected with a patient reported outcome questionnaire
Symptoms experienced during defecation | Ten weeks after inclusion
  Symptoms experienced during defecation will be collected with a patient reported outcome questionnaire
Symptoms experienced during defecation | Twenty-four weeks after inclusion
  Symptoms experienced during defecation will be collected with a patient reported outcome questionnaire
Frequency of digital help during defecation | Ten weeks after inclusion
  The frequency of digital stimulation will be collected with a patient reported outcome questionnaire
Frequency of digital help during defecation | Twenty-four weeks after inclusion
  The frequency of digital stimulation will be collected with a patient reported outcome questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Siproudhis, Md, PhD, Principal Investigator — Rennes University Hospital
Locations (6):
- France (6):
  - CHRU de Lille, Lille
  - CHU de Nantes, Nantes
  - CMRRF de Kerpape, Ploemeur
  - Rennes University Hospital, Rennes
  - CHU de Rouen, Rouen
  - CHRU de Nancy-Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Brochard C, Jezequel M, Blanchard-Dauphin A, Kerdraon J, Perrouin-Verbe B, Leroi AM, Reymann JM, Peyronnet B, Morcet J, Siproudhis L. Transanal irrigation is a better choice for bowel dysfunction in adults with Spina bifida: A randomised controlled trial. Colorectal Dis. 2023 Jun;25(6):1267-1276. doi: 10.1111/codi.16518. Epub 2023 Mar 11. PMID 36799340